CLINICAL TRIAL: NCT00281983
Title: Pilot Study on Allogeneic Stem Cell Transplantation Following Conditioning With Fludarabine and an Alkylating Agent in Patients With High-Risk Chronic Lymphocytic Leukemia
Brief Title: Fludarabine and Cyclophosphamide in Treating Patients Who Are Undergoing Donor Stem Cell Transplant for Chronic Lymphocytic Leukemia or Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL3X; EU-20554; MEDAC-FLUD.10/CLL
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2007-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; Waldenström macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab; Antilymphocyte Serum; Filgrastim; Rituximab; Busulfan; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

ARMS (1):
- Allogeneic stem cell transplantation (Experimental): 1. Cytoreductive therapy for inducing a state of partial remission:
     FC or FC-R or alternative salvage regimens (e.g. Alemtuzumab)
  2. Conditioning regimen:
     FC +/- ATG (Arm A) or FC/Busulfan +/- ATG (Arm C: refractory patients only)
  3. allogeneic-PBSCT (from HLA-identical donor)
  4. GVHD prophylaxis: CSA + MTX or MMF
  5. +/- DLI (Donor lymphocyte infusions)
  Interventions: Biological: alemtuzumab; Biological: anti-thymocyte globulin; Biological: filgrastim; Biological: rituximab; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: alemtuzumab
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: rituximab
Biological: therapeutic allogeneic lymphocytes
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as alemtuzumab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving methotrexate, cyclosporine and mycophenolate mofetil after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

PURPOSE: This phase I/II trial is studying the side effects of giving fludarabine together with cyclophosphamide and to see how well they work in treating patients who are undergoing donor stem cell transplant for B-cell chronic lymphocytic leukemia or Waldenström's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and safety of induction therapy comprising fludarabine and cyclophosphamide followed by allogeneic stem cell transplantation in patients with high-risk B-cell chronic lymphocytic leukemia or lymphoplasmocytic lymphoma (Waldenstrom's macroglobulinemia).

Secondary

* Determine the incidence and kinetics of clinical and molecular remissions in patients treated with this regimen.
* Determine event-free and overall survival of patients treated with this regimen.
* Determine the duration of clinical and molecular remission in relation to the underlying cytogenetic deviation in patients treated with this regimen.
* Determine the kinetics and extent of lympho-hematopoietic donor chimerism in patients treated with this regimen.

OUTLINE: This is a multicenter, open-label, nonrandomized, pilot study.

* Cytoreductive therapy: Patients receive up to 3 courses of cytoreductive therapy comprising fludarabine IV and cyclophosphamide IV on days 1-3 (with or without rituximab IV on day 1). Patients refractory to fludarabine-containing therapy may receive alemtuzumab IV for 12 weeks OR any other cytotoxic salvage regimen for cytoreduction.
* Conditioning regimen: Patients receive 1 of the following conditioning regimens*:

NOTE: *Patients who did not achieve partial response after cytoreductive therapy receive regimen 3.

* Regimen 1: Patients receive fludarabine IV and cyclophosphamide IV on days -7 to -3. If stem cells are collected from an unrelated donor, patients also receive anti-thymocyte globulin (ATG) IV on days -4 to -1.
* Regimen 2: Patients undergo total-body irradiation on day -9. Patients then receive alemtuzumab IV on days -8 to -4 and fludarabine IV and cyclophosphamide IV on days -6 to -2.
* Regimen 3: Patients receive fludarabine IV on days -7 to -3, busulfan IV or orally on days -7 to -5, and cyclophosphamide IV on days -3 to -2. If stem cells are collected from an unrelated donor, patients also receive ATG on days -3 to -1.

  * Allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo allogeneic PBSCT on day 0. Patients receive filgrastim (G-CSF) subcutaneously daily starting on day 5 and continuing until blood count recover.
  * Graft-versus-host-disease (GVHD) prophylaxis: Patients receive cyclosporine IV beginning on day -1 and continuing until approximately day 100. Patients treated with conditioning regimen 1 or 3 also receive methotrexate IV on days 1, 3, and 6 OR oral mycophenolate mofetil twice daily on days 0-50. Patients with evidence of residual disease at least 4 weeks after completion of cyclosporine undergo donor lymphocyte infusion (DLI).
  * DLI: The donor T-lymphocytes are collected from the PBSCT donor without prior G-CSF mobilization. Patients receive DLI every 8 weeks in the presence of residual disease and the absence of GVHD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia or lymphoplasmocytic lymphoma (Waldenstrom's macroglobulinemia)

  * Must have poor prognostic features and low probability of successful autografting, defined by one of the following criteria:

    * Progressive disease with unfavorable cytogenetics (deletion or mutation of critical regions on chromosomes 11q and/or 17p [p53]; and/or unmutated status of the immunoglobulin V_H gene region; and/or usage of the V_H 3-21 gene), defined as 1 of the following:

      * Doubling of lymphocyte count or nodal involvement within 3 months or less
      * Progressive decline of platelet count and/or hemoglobin values defining Binet stage C disease (or to 50% or less of baseline values within 3 months) not due to immune mechanisms
      * Symptomatic splenomegaly
      * Discomfort or imminent complications due to large tumor masses
      * B symptoms
    * Refractory disease or early relapse (within 12 months) after treatment with a fludarabine-containing regimen
    * Relapsed after autologous stem cell transplant (SCT)
    * Insufficient stem cell harvest for intended autologous SCT
* Presence of a clonal CDR III rearrangement detected by polymerase chain reaction
* No Richter's syndrome
* HLA-identical sibling or unrelated donor available

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 1
* Creatinine clearance > 60 mL/min
* SGOT, SGPT, and bilirubin < 2 times normal
* Normal cardiac function determined by ECG and echocardiographic examination
* Inspiratory vital capacity, FEV_1, and DLCO > 50% of predicted
* No serious localized or systemic infections
* No other concurrent malignant disease
* No impaired organ function
* No uncontrolled diabetes
* No uncontrolled hypertension
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No HIV infection
* No hepatitis B or C infection
* No concurrent alcohol or drug abuse
* No dementia or altered mental status that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-06; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the proportion of eligible patients completing the transplant procedure successfully
Safety as measured by a treatment-related mortality of < 25% at 2 years following transplant

SECONDARY OUTCOMES:
Clinical remission rate by NIH criteria at 12 months following transplant
Minimal residual disease negativity rate as measured by high-resolution flow or CDR PCR at 12 months following transplant
Chimerism as measured by STR-PCR at 12 months following transplant
Event-free and overall survival at 5 years following transplant

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dreger, Study Chair — Universitaets-Kinderklinik Heidelberg
Locations (13):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada
- Germany (12):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Goettingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - University Hospital of Leipzig, Leipzig
  - Klinikum der Universitaet Regensburg, Regensburg
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dreger P, Dohner H, Ritgen M, Bottcher S, Busch R, Dietrich S, Bunjes D, Cohen S, Schubert J, Hegenbart U, Beelen D, Zeis M, Stadler M, Hasenkamp J, Uharek L, Scheid C, Humpe A, Zenz T, Winkler D, Hallek M, Kneba M, Schmitz N, Stilgenbauer S; German CLL Study Group. Allogeneic stem cell transplantation provides durable disease control in poor-risk chronic lymphocytic leukemia: long-term clinical and MRD results of the German CLL Study Group CLL3X trial. Blood. 2010 Oct 7;116(14):2438-47. doi: 10.1182/blood-2010-03-275420. Epub 2010 Jul 1. PMID 20595516
- [Result] Ritgen M, Bottcher S, Stilgenbauer S, Bunjes D, Schubert J, Cohen S, Humpe A, Hallek M, Kneba M, Schmitz N, Dohner H, Dreger P; German CLL Study Group. Quantitative MRD monitoring identifies distinct GVL response patterns after allogeneic stem cell transplantation for chronic lymphocytic leukemia: results from the GCLLSG CLL3X trial. Leukemia. 2008 Jul;22(7):1377-86. doi: 10.1038/leu.2008.96. Epub 2008 Apr 17. PMID 18418404
- [Result] Dreger P, Schnaiter A, Zenz T, Bottcher S, Rossi M, Paschka P, Buhler A, Dietrich S, Busch R, Ritgen M, Bunjes D, Zeis M, Stadler M, Uharek L, Scheid C, Hegenbart U, Hallek M, Kneba M, Schmitz N, Dohner H, Stilgenbauer S. TP53, SF3B1, and NOTCH1 mutations and outcome of allotransplantation for chronic lymphocytic leukemia: six-year follow-up of the GCLLSG CLL3X trial. Blood. 2013 Apr 18;121(16):3284-8. doi: 10.1182/blood-2012-11-469627. Epub 2013 Feb 22. PMID 23435461
- [Result] Scheffold A, Jebaraj BMC, Jaramillo S, Tausch E, Steinbrecher D, Hahn M, Bottcher S, Ritgen M, Bunjes D, Zeis M, Stadler M, Uharek L, Scheid C, Hegenbart U, Hallek M, Kneba M, Schmitz N, Dohner H, Dreger P, Stilgenbauer S. Impact of telomere length on the outcome of allogeneic stem cell transplantation for poor-risk chronic lymphocytic leukaemia: results from the GCLLSG CLL3X trial. Br J Haematol. 2017 Oct;179(2):342-346. doi: 10.1111/bjh.14219. Epub 2016 Jul 8. No abstract available. PMID 27391907
- [Result] Kramer I, Stilgenbauer S, Dietrich S, Bottcher S, Zeis M, Stadler M, Bittenbring J, Uharek L, Scheid C, Hegenbart U, Ho A, Hallek M, Kneba M, Schmitz N, Dohner H, Dreger P. Allogeneic hematopoietic cell transplantation for high-risk CLL: 10-year follow-up of the GCLLSG CLL3X trial. Blood. 2017 Sep 21;130(12):1477-1480. doi: 10.1182/blood-2017-04-775841. Epub 2017 Jul 17. No abstract available. PMID 28716861